CLINICAL TRIAL: NCT06451029
Title: Integrated Primary and Secondary Prevention of Smoking Related Diseases With Low Dose CT Scan and Circulating Biomarkers, Coupled With Personalised Smoking Cessation Activity
Brief Title: Prevention of Smoking Related Diseases
Acronym: LSP-3
Status: Recruiting | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Pierluigi Novellis, Medical Doctor, Scientific Institute San Raffaele
Other Study IDs: 136/INT/2021
Record Dates: First submitted 2024-05-30; First posted 2024-06-10 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer; Lung Cancer Screening; Smoking Cessation
Keywords: lung cancer screening; smoking cessation; counseling
MeSH Terms: conditions — Lung Neoplasms; Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- face-to-face interviews: The group that will carry out the psychological counselling in the presence will have 6 meetings (spread over 6 months) with a psychologist at the anti-smoking center in the hospital and a final phone call 12 months after the first meeting to verify the maintenance of abstinence.
- video interviews: The group that will be followed in remote mode will carry out the same number of interviews as the group described above and a 12-months call will also be made to them to check the state of abstinence.

SUMMARY:
This is a prospective, observational, monocentric study. This study wants to test if among a smoking cessation intervention, behavioural counselling by video session is related to higher compliance and higher success rate than standard smoking cessation activity (face to face counselling).

DETAILED DESCRIPTION:
This intervention was structured on Sitab guidelines (Società Italiana Tabaccologia - Italian Tobacco Society), who suggest to use long-term counseling for at least six months and preferably for 12, in order to strengthen abstinence and cover the period with the highest risk of relapse. Clinicians who follow these guidelines must provide a path greater than or equal to 4 meetings and they will have a greater degree of success if the time that will be devoted to meetings is consistent. The group that will carry out the psychological counselling in the presence will have 6 meetings (spread over 6 months) with a psychologist at the anti-smoking center of the San Raffaele Hospital and a final phone call 12 months after the first meeting to verify the maintenance of abstinence. The meetings at the anti-smoking center are aimed at monitoring the progress of the smoking cessation process, thanks also to tests (fagestrom test, motivational questionnaire, smoker's diary) and prevent any drop outs. The group that will be followed in remote mode will carry out the same number of interviews as the group described above and a 12-months call will also be made to them to check the state of abstinence. The difference between the two groups is in the way interviews were conducted.

Both face-to-face interviews and those through videocall allow smokers, in addition to learning strategies to limit the consumption of the substance, to share the path towards de-exhaustion with a professional and be supported by it.

The subdivision into the two groups will be carried out through voluntary choice of participants.

ELIGIBILITY:
Inclusion Criteria:

* Strong smokers (pack years >= 20)
* Over or equal the age of 50
* Able to sign specific informed consent for the study

Exclusion Criteria:

* Not having plans to quit smoking

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Strong smokers enrolled in the lung cancer screening program.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Create an innovative smoking cessation program with personalized and tailored primary prevention support within screening programs. | from enrollment to the end treatment at 1 year
  The study aims to evaluate the difference in success between standard anti-smoking psychological counselling, conducted through face-to-face interviews, and anti-smoking psychological counselling conducted through remote video interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Institute Ospedale San Raffaele, Milan, Italy, Milan, Italy

IPD SHARING:
Plan to Share IPD: No